CLINICAL TRIAL: NCT02412189
Title: Pressure-dependent Changes in Hematocrit and Plasma Volume During Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Tor Damén, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TDamen
Record Dates: First submitted 2015-03-10; First posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Blood Pressure; Hematocrit Change; Anesthesia
Keywords: Anesthesia; Blood pressure; Plasma volume; Vasopressor agents; Continuous noninvasive hemoglobin measurement; Coronary artery bypass
MeSH Terms: interventions — Norepinephrine; Vasoconstrictor Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): Ordinary anesthesia, mean arterial pressure allowed to decrease to 60 mmHg. If it is lower the patients will receive a norepinephrine infusion in order to raise the mean arterial pressure to 60 mmHg.
- Maintained blood pressure (Active Comparator): Ordinary anaesthesia and maintained preanesthetic blood pressure by norepinephrine infusion
  Interventions: Procedure: Maintained blood pressure; Drug: Norepinephrine

INTERVENTIONS:
Procedure: Maintained blood pressure — Norepinephrine therapy to maintain preanesthesia blood pressure
  Arms: Maintained blood pressure
Drug: Norepinephrine — Norepinephrine therapy to maintain preanesthesia blood pressure
  Other Names: Vasopressor
  Arms: Maintained blood pressure

SUMMARY:
The arterial blood pressure affects the ratio between filtration and reabsorption of fluids in the circulating blood volume and thereby the hematocrit. During induction of anesthesia blood pressure, hemoglobin level and hematocrit decreases. The aim of the study is to evaluate weather a maintained blood pressure with norepinephrine during anesthesia induction reduces the decrease in hematocrit.

DETAILED DESCRIPTION:
24 patients scheduled for coronary artery bypass surgery will be included and randomized to receive either norepinephrine in the dose needed to maintain pre-anesthesia blood pressure or to a control group and receive norepinephrine only if mean arterial pressure decreases below 60 mmHg. Arterial blood gas will be analysed every ten minutes. Equal anesthesia in both groups will be monitored. No fluids will be infused. Noninvasive continuous hemoglobin measurement (SpHb) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Elective coronary artery surgery patients

Exclusion Criteria:

* Age under 18 years
* untreated hypertension
* a reduced left ventricular systolic ejection fraction of 45 % or less
* diabetes mellitus
* former stroke and/or a known carotid artery stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-04 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
The magnitude and dynamics of the decrease in hematocrit during anesthesia induction | 70 minutes from anesthesia induction

SECONDARY OUTCOMES:
Reduced hematocrit decrease by vasopressor infusion maintained blood pressure | 70 minutes from anesthesia induction
  To assess if the decrease in hematocrit can be reduced, by maintaining the blood pressure with vasopressor infusion

OTHER OUTCOMES:
Accuracy of continuous non-invasive hemoglobin monitoring (SpHb) to invasive Hb levels | 70 minutes from anesthesia induction
  To evaluate if changes in invasive measured Hb levels, can be measured by continuous non-invasive hemoglobin monitoring (SpHb).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nygren, MD PHD, Principal Investigator — Sweden: Sahlgrenska University hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden, Sweden